CLINICAL TRIAL: NCT03263923
Title: GIFT Web Based Resourcefulness Training for Grandmother Caregivers
Brief Title: The Grandmother Study: Grandmother Initiatives in Family Transformation
Acronym: GIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Carol M. Musil, Principal Investigator, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01NR015999 (NIH)
Record Dates: First submitted 2017-08-21; First posted 2017-08-28 (Actual); Results first posted 2022-10-12 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Women; Grandmother
Keywords: grandmother caregivers; grandfamily; grandfamilies; custodial grandparent; custodial grandmother; multigenerational family; Grandmothers raising or living with grandchildren

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Who Masked: Participant
Masking Description: Participants randomly assigned to groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Cognitive behavioral skills training & 4 wks online journaling (Experimental): Cognitive behavioral skills' training and 4 weeks of online journaling.
  Participants receive cognitive behavioral skills training by online video, then participants must complete a 28 day online journal reflecting on the cognitive skills they used to handle various situations.
  Interventions: Behavioral: Cognitive behavioral intervention and journaling
- Arm 2: Reflective journaling training & 4 wks online journaling (Active Comparator): Reflective journaling training and 4 weeks of online journaling.
  Participants watch a reflective journaling video and complete a 28 day journal using a different set of prompts to reflect on their days and describe how they handled various situations.
  Interventions: Behavioral: Reflective journaling

INTERVENTIONS:
Behavioral: Cognitive behavioral intervention and journaling — Cognitive behavioral skills training and 4 weeks of online journaling
  Arms: Arm 1: Cognitive behavioral skills training & 4 wks online journaling
Behavioral: Reflective journaling — Reflective journaling training and 4 weeks of online journaling
  Training in reflective journaling and 4 weeks of online journaling
  Arms: Arm 2: Reflective journaling training & 4 wks online journaling

SUMMARY:
CWRU Research Study: Looking for grandmothers living with grandchildren, 18 years of age or younger, to take part in a study to compare methods of dealing with the stress of caregiving to grandchildren. Participants need to have daily access to a computer, complete four surveys online, and be willing to write in a journal every day for a month. Participants will be compensated for their time.

DETAILED DESCRIPTION:
This is a randomized clinical trial that will compare two methods of dealing with stress of grandparent caregiving to grandchildren.

ELIGIBILITY:
Inclusion Criteria:

* Grandmother to one or more grandchildren (age 18 or younger) living in the same home (with or without parents)

Exclusion Criteria:

1. Grandmothers to grandchildren who do not share their home
2. Not a grandmother
3. Not living in the United States.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — female
Enrollment: 346 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol M Musil, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- CWRU, Cleveland, Ohio, United States

REFERENCES:
- [Result] Wallace MK, Still CH, Jeanblanc AB, Musil CM. Successful and Cost-Effective Facebook Recruitment: Is It Possible? Results From a Longitudinal Randomized Clinical Trial in Grandmother Caregivers. Int J Aging Hum Dev. 2021 Dec;93(4):1031-1050. doi: 10.1177/0091415020987667. Epub 2021 Feb 17. PMID 33593072
- [Result] Tracy EM, Braxton R, Henrich C, Jeanblanc A, Wallace M, Burant CJ, Musil C. Grandmothers raising grandchildren: managing, balancing and maintaining family relationships. J Women Aging. 2022 Nov-Dec;34(6):757-772. doi: 10.1080/08952841.2021.1951114. Epub 2021 Jul 15. PMID 34265228
- [Result] Musil CM, Wallace MK, Jeanblanc AB, Toly VB, Zauszniewski JA, Burant CJ. Theoretical and Operational Consideration of Mindfulness, Resilience, and Resourcefulness. West J Nurs Res. 2021 Mar;43(3):210-218. doi: 10.1177/0193945920956684. Epub 2020 Sep 3. PMID 32880239
- [Result] Wallace MK, Jeanblanc AB, Musil CM. Incidental findings: A practical protocol for reporting elevated depressive symptoms in behavioral health research. Arch Psychiatr Nurs. 2020 Jun;34(3):96-99. doi: 10.1016/j.apnu.2020.04.005. Epub 2020 Apr 13. PMID 32513473
- [Result] Dolbin-MacNab ML, Jeanblanc AB, Musil CM, Infurna FJ, Smith GC. Supporting grandchildren's remote instruction during COVID-19: Experiences of custodial grandmothers. Psychol Sch. 2022 Apr 29:10.1002/pits.22714. doi: 10.1002/pits.22714. Online ahead of print. PMID 35572175

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Cognitive Behavioral Skills Training & 4 Wks Online Journaling | Arm 2: Reflective Journaling Training & 4 Wks Online Journaling
Started (Enrolled, consented, Participants who were sent the baseline questionnaire.) | 174 | 172
Completed Enrolled Participants Who Completed the Baseline Questionnaire | 173 | 169
Completed Intervention and T2 Questionnaire | 149 | 151
Completed | 149 | 151
Not Completed | 25 | 21
Not completed — Withdrawal by Subject | 10 | 8
Not completed — Lost to Follow-up | 15 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Cognitive Behavioral Skills Training & 4 Wks Online Journaling | Arm 2: Reflective Journaling Training & 4 Wks Online Journaling | Total
Number analyzed (Participants) | 173 | 169 | 342
Age, Continuous [Mean (Standard Deviation); unit: years] — Age, reported in years, at baseline
  years | 55.792 (7.080) | 56.584 (8.052) | 56.194 (7.588)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender was not directly measured. Participants were eligible for enrollment if they self-identified as a "grandmother" living with grandchildren.
  Participants
    Female | 173 | 169 | 342
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Participants were asked (yes/no) whether they identified as Hispanic or Latina. Asked separately from race.
  Participants
    Hispanic or Latino | 12 | 17 | 29
    Not Hispanic or Latino | 161 | 152 | 313
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Participants were asked to select their preferred racial identity from the list given here. Participants could select as many as applied and also had the option to select "other" or "prefer not to answer.
  Participants
    Self-identified racial identity: American Indian or Alaska Native | 1 | 1 | 2
    Self-identified racial identity: Asian | 1 | 0 | 1
    Self-identified racial identity: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Self-identified racial identity: Black or African American | 30 | 34 | 64
    Self-identified racial identity: White | 124 | 122 | 246
    Self-identified racial identity: More than one race | 8 | 5 | 13
    Self-identified racial identity: Unknown or Not Reported | 9 | 7 | 16
Region of Enrollment [Number; unit: participants]
  United States | 173 | 169 | 342
Marital Status [Count of Participants; unit: Participants] — Participants asked their current domestic arrangements. Responses collapsed into a dichotomous measure of Married/Living with a Partner or Single
  Participants
    Married or living with a partner | 86 | 84 | 170
    Not married or living with a partner | 87 | 85 | 172
Job Status [Count of Participants; unit: Participants] — Participants asked whether they were employed in a paying job
  Participants
    Working full-time | 63 | 54 | 117
    Working part-time | 20 | 30 | 50
    Not working | 90 | 85 | 175
Educational Attainment [Count of Participants; unit: Participants] — Participants were asked "How far did you go in school?"
  Participants
    8 years or less | 1 | 1 | 2
    Some high school | 2 | 6 | 8
    High school complete/GED | 26 | 31 | 57
    Post high school, business or trade school | 19 | 13 | 32
    1-3 years of college, no degree completed | 45 | 47 | 92
    Completed Associate's or other 2 year degree | 31 | 28 | 59
    4 years college (completed degree) | 30 | 24 | 54
    Graduate school | 19 | 19 | 38
Number of co-residential grandchildren [Count of Participants; unit: Participants] — Participants were asked how many of their grandchildren live with them on a daily basis.
  Participants
    One (1) in-home grandchild | 93 | 75 | 168
    Two (2) in-home grandchildren | 45 | 57 | 102
    Three (3) in-home grandchildren | 21 | 26 | 47
    Four (4) in-home grandchildren | 11 | 6 | 17
    Five (5) in-home grandchildren | 3 | 3 | 6
    Six (6) in-home grandchildren | 0 | 1 | 1
    Seven (7) in-home grandchildren | 0 | 1 | 1
Self-appraised caregiving stress [Mean (Standard Deviation); unit: score on scale] — Participants were asked to rate their stress associated with living with and raising grandchildren on a continuous sliding scale from 0-10 (0=no stress).
  score on scale | 7.847 (2.394) | 7.131 (2.575) | 7.419 (2.410)
Self-appraised caregiving reward [Mean (Standard Deviation); unit: score on scale] — Participants were asked to rate the amount of reward they feel associated with living with and raising grandchildren on a continuous sliding scale from 0-10 (0=no reward).
  score on scale | 7.865 (2.43) | 7.847 (2.394) | 7.856 (2.410)
Duke Subjective Social Support [Mean (Standard Deviation); unit: score on scale] — Composite score representing the amount of subjective social support participants receive from family and friends. Derived from the Subjective Social Support subscale items of the Duke Social Support Index. Scores range from 0-14, higher scores indicate more support.
  score on scale | 8.775 (3.236) | 8.773 (3.443) | 8.774 (3.338)
Duke Instrumental Social Support [Mean (Standard Deviation); unit: score on scale] — Composite score representing the amount of instrumental social support participants receive from family and friends. Derived from the Instrumental Social Support subscale items of the Duke Social Support Index. Scores range from 0-13, higher scores indicate more support.
  score on scale | 5.965 (3.443) | 5.799 (3.236) | 5.883 (3.338)
Resourcefulness [Mean (Standard Deviation); unit: score on scale] — Composite measure of Resourcefulness, from the 28 items of Zausniewski et al's Resourcefulness scale. Possible scores range from 0-140, higher scores represent greater resourcefulness.
  score on scale | 81.208 (19.237) | 81.630 (18.079) | 81.422 (18.631)
Depressive Cognitions [Mean (Standard Deviation); unit: score on scale] — Composite scale capturing negative thinking patterns that precede clinical depression. comprising of items from Zausniewski's Depressive Cognitions Scale. Possible scores range from 0-40, higher scores reflect more depressive cognitions
  score on scale | 7.799 (5.592) | 7.76 (6.09) | 7.781 (5.841)
Caregiving status [Count of Participants; unit: Participants]
  Primary caregivers (grandchild(ren), no parents live with grandmother) | 143 | 140 | 283
  Multigenerational caregivers (grandchild(ren) and at least 1 parent live with grandmother) | 30 | 29 | 59
Intra-family strain [Mean (Standard Deviation); unit: score on scale] — Intra-family strain was assessed with a 10- item composite scale of the intra-family strain subscale of the Family Inventory of Life Events (FILE) (McCubbin, et al., 1996). Participants response to 10 yes/no questions about stressful events that may have happened in their family. Scores range from 0-10 and higher scores represent more strain.
  score on scale | 5.256 (2.460) | 5.107 (2.570) | 5.182 (2.513)
Family income [Count of Participants; unit: Participants] — Participants were asked to select the category their monthly household income fit into.
  Participants
    Under $999/month | 16 | 20 | 36
    $1,000-2,000/month | 32 | 41 | 73
    $2,001-3,000/month | 32 | 27 | 59
    $3,001-4,000/month | 18 | 26 | 44
    $4,001-5,000/month | 22 | 24 | 46
    Over $5,000/month | 37 | 23 | 60
    Prefer not to answer | 16 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Depressive Symptoms
Description: Center for Epidemiologic Disease - Depression Scale (CES-D) Radloff, 1977. Composite item derived from 20 item scale. Individual items are scored on a 4 point likert scale (0-3). Individual items are summed and possible scale scores range from 0-60. Higher scores represent greater depressive symptoms. Scores of 16 or greater are interpreted as indicating an increased risk of diagnosis of clinical depression.
Time Frame: comparison of baseline with 24 weeks post journaling completion
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Arm 1: Cognitive Behavioral Skills Training & 4 Wks Online Journaling (N=149): Cognitive behavioral skills' training and 4 weeks of online journaling.
  Participants receive cognitive behavioral skills training by online video, then participants must complete a 28 day online journal reflecting on the cognitive skills they used to handle various situations.
- Arm 2: Reflective Journaling Training & 4 Wks Online Journaling (N = 151): Reflective journaling training and 4 weeks of online journaling.
  Participants watch a reflective journaling video and complete a 28 day journal using a different set of prompts to reflect on their days and describe how they handled various situations.
Arm/Group | Arm 1: Cognitive Behavioral Skills Training & 4 Wks Online Journaling (N=149) | Arm 2: Reflective Journaling Training & 4 Wks Online Journaling (N = 151)
Number analyzed (Participants) | 149 | 151
score on a scale
  Time 1 (baseline) | 18.116 (11.650) | 18.231 (11.51)
  Time 4 (24 wks post-journaling) | 15.135 (11.650) | 15.873 (10.425)

2. Primary Outcome: Well Being
Description: SF 12 individual item: overall self-appraised health. This is a single response item "In general, would you say your health is..." Participants respond on 5 point scale with response options ranging from Poor (1) to Excellent (5). Higher scores indicate better self-appraised health.
Time Frame: comparison of baseline with 24 weeks post journaling
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Cognitive Behavioral Skills Training & 4 Wks Online Journaling (N=149) | Arm 2: Reflective Journaling Training & 4 Wks Online Journaling (N = 151)
Number analyzed (Participants) | 149 | 151
score on a scale
  Time 1 (baseline) | 2.97 (.974) | 3.00 (.982)
  Time 4 (24 wks post-journaling) | 2.92 (.929) | 2.95 (.909)

3. Primary Outcome: Family Well Being - Composite Score Derived From 12 Items.
Description: General Family Functioning 12 item subscale of the McMaster Family Assessment Device (FAD). Participants respond on a 5 point likert scale. The subscale is the mean of the participant's responses to the 12 items with possible composite scores of 0-5. Higher scores indicate worse family well being.
Time Frame: comparison of baseline with 24 weeks post journaling
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Cognitive Behavioral Skills Training & 4 Wks Online Journaling (N=149) | Arm 2: Reflective Journaling Training & 4 Wks Online Journaling (N = 151)
Number analyzed (Participants) | 149 | 151
score on a scale
  Time 1 (baseline) | 2.300 (.532) | 2.300 (.503)
  Time 4 (24 wks post-journaling) | 2.172 (.600) | 2.172 (.564)

4. Primary Outcome: SF-12 Mental Health Composite Score
Description: Normed score generated by vendor-provided software using all 12 items of the SF-12v2 Health Survey. Scores range from 0-100, with higher scores indicating better mental health.
  Note: the SF-12 measures 8 health domains (Physical Function, Bodily Pain, Vitality, Role-Emotional, Role-Physical, General Health, Social Function, Mental Health) across 12 individual response questions. All 12 responses are normed for gender, and country of origin and differentially weighted to calculate scores for both physical and mental health.
Time Frame: Baseline vs 24 week followup
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Arm 1: Cognitive Behavioral Skills Training & 4 Wks Online Journaling: Cognitive behavioral skills' training and 4 weeks of online journaling.
  Participants receive cognitive behavioral skills training by online video, then participants must complete a 28 day online journal reflecting on the cognitive skills they used to handle various situations.
  Cognitive behavioral intervention and journaling: Cognitive behavioral skills training and 4 weeks of online journaling
- Arm 2: Reflective Journaling Training & 4 Wks Online Journaling: Reflective journaling training and 4 weeks of online journaling.
  Participants watch a reflective journaling video and complete a 28 day journal using a different set of prompts to reflect on their days and describe how they handled various situations.
  Reflective journaling: Reflective journaling training and 4 weeks of online journaling
  Training in reflective journaling and 4 weeks of online journaling
Arm/Group | Arm 1: Cognitive Behavioral Skills Training & 4 Wks Online Journaling | Arm 2: Reflective Journaling Training & 4 Wks Online Journaling
Number analyzed (Participants) | 149 | 151
score on a scale
  T1 (baseline) | 43.452 (11.298) | 41.613 (12.003)
  T4 (24 week followup post journal) | 45.611 (11.001) | 45.230 (10.357)

5. Primary Outcome: SF-12 Physical Health Composite Score
Description: Normed score generated by vendor-provided software using all 12 items of the SF-12v2 Health Survey. Scores range from 0-100, with higher scores indicating better physical health.
  Note: the SF-12 measures 8 health domains (Physical Function, Bodily Pain, Vitality, Role-Emotional, Role-Physical, General Health, Social Function, Mental Health) across 12 individual response questions. All 12 responses are normed for gender, and country of origin and differentially weighted to calculate scores for both physical and mental health.
Time Frame: Baseline vs 24 week followup
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Cognitive Behavioral Skills Training & 4 Wks Online Journaling | Arm 2: Reflective Journaling Training & 4 Wks Online Journaling
Number analyzed (Participants) | 149 | 151
score on a scale
  T1 (Baseline) | 44.344 (11.907) | 45.125 (11.700)
  T4 (24 week followup post journal) | 44.654 (11.303) | 44.506 (11.531)

ADVERSE EVENTS:
Time Frame: Participants were screened for depressive symptoms (using the CES-D 20 item scale) at baseline (T1) and 2 weeks (T2), 12 weeks (T3), and 24 weeks post-intervention (T4).
Arm/Group | Arm 1: Cognitive Behavioral Skills Training & 4 Wks Online Journaling | Arm 2: Reflective Journaling Training & 4 Wks Online Journaling
All-Cause Mortality (participants affected / at risk) | 0/173 | 0/169
Serious Adverse Events (participants affected / at risk) | 0/173 | 0/169
Other Adverse Events (participants affected / at risk) | 52/173 | 45/169
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Cognitive Behavioral Skills Training & 4 Wks Online Journaling (N=173) | Arm 2: Reflective Journaling Training & 4 Wks Online Journaling (N=169)
Elevated depressive symptoms at T1: Baseline (Psychiatric disorders) | 31 (31) | 31 (31) — CES-D scores over 30
Elevated depressive symptoms at T2: 2 weeks post-intervention (Psychiatric disorders) | 9 (9) | 9 (9)
Elevated depressive symptoms at T3: 12 weeks post-intervention (Psychiatric disorders) | 13 (13) | 17 (17)
Elevated depressive symptoms at T4: 24 weeks post-intervention (Psychiatric disorders) | 8 (8) | 13 (13)

LIMITATIONS AND CAVEATS:
Does not include grandfathers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/23/NCT03263923/Prot_SAP_000.pdf